CLINICAL TRIAL: NCT02671097
Title: A Phase 1, Open Label, Fixed-sequence Study to Evaluate the Effect of BAY1841788 (ODM-201) on Drug Transporters Using Rosuvastatin as Probe Substrate and to Assess Pharmacokinetics and Safety of BAY1841788 in Female and Male Volunteers
Brief Title: Drug-drug Interaction Study Using Rosuvastatin as a Breast Cancer Resistant Protein (Efflux Transporter), Organic Anion-transporting Polypeptide (OATP)1B1, and OATP1B3 (Uptake Transporters) Probe Substrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 17723; 2015-003244-38 (EudraCT Number)
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Volunteers; Pharmacokinetics; Drug Interaction
MeSH Terms: interventions — Rosuvastatin Calcium; darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BAY1841788 (ODM-201) + Rosuvastatin (Experimental): All subjects will receive a single dose BAY1841788 (ODM-201) (600 mg) followed by multiple doses BAY1841788 (ODM-201) (600 mg BID) as well as 2 times a single dose rosuvastatin (5 mg), once alone and once in combination with BAY1841788 (ODM-201).
  Interventions: Drug: Rosuvastatin; Drug: BAY1841788 (ODM-201)

INTERVENTIONS:
Drug: Rosuvastatin — 5 mg tablet single dose on Day 01 in Period 1 and on Day 08 in Period 2.
Drug: BAY1841788 (ODM-201) — 600 mg single dose, administered as 2 x 300 mg tablets on Day 01 in Period 2; 600 mg BID multiple dose, administered as 2 x 300 mg tablets on Day 04 to Day 08 in Period 2.

SUMMARY:
Evaluation of the potential perpetrator effect of BAY1841788 (ODM-201) on rosuvastatin pharmacokinetics.

PK of BAY1841788 (ODM-201) after single and repeated administration in male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject - as determined by medical history, physical examination and all procedures required by this protocol.
* Age: 45 to 65 years at the screening visit.
* Race: White.
* Body mass index (BMI): ≥18.0 and ≤29.9 kg/m*2.
* Adequate venous access (frequent blood sampling).
* Ability to understand and follow study-related instructions.
* Females have to be in postmenopausal state, revealed by: Medical history, if applicable (natural menopause at least 12 months prior to first study drug administration; or surgical menopause by bilateral ovariectomy at least 3 months prior to first study drugadministration) and follicle stimulating hormone (FSH) >40 IU/L at screening examination.
* Male subjects must agree to use condoms as an effective contraception barrier method during the whole study (starting after informed consent) and for 3 months after the end of treatment with BAY1841788 (ODM-201). In addition, participants must agree to utilize a second reliable method of contraception simultaneously. The second method which has to be used by a female partner of childbearing potential can be one of the following methods: diaphragm or cervical cap with spermicide or intra-uterine device or hormone-based contraception.

Exclusion Criteria:

* Medical and surgical history

  * Subjects with clinically relevant findings in medical history e.g. history or currently existing relevant diseases of vital organs, central nervous system (for example seizures) or other organs (e.g. diabetes mellitus).
  * Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
  * Febrile illness within 1 week before the first study drug administration.
  * A medical history of risk factors for Torsades de Pointes (e.g. family history of Long QT interval in electrocardiogram Syndrome) or other arrhythmias.
* History of myopathia after treatment with statins.

  * History of rhabdomyolysis or myopathia.
  * Medical history of any type of psychiatric disorder, especially mood disorders including medical history with suicidal ideation and/or suicide attempts.
  * History of thyroid disorders, especially hypothyreosis.
  * History of respiratory disorder (excluding history of bronchitis or pneumonia).
  * History of myasthenia.
  * History of muscle pain or muscle ache, muscle soreness of unknown origin or on frequent occasions although an origin might have been found.
  * History of any clinically significant hypoglycemia or hyperglycemia.
  * Relevant hepatic disorders like a history of viral hepatitis, cholestasis, disturbances of bilirubin metabolism, any progressive liver disease.
  * Relevant renal disorders like recurrent glomerulonephritis, renal injury, and renal insufficiency. However, a history of a single episode of uncomplicated nephrolithiasis will not prevent participation.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of Rosuvastatin from time zero to 24 hours (AUC(0-24)) | Before Rosuvastatin administration, as well as 30 min, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 h after Rosuvastatin administration
Maximum drug concentration (Cmax) in plasma of Rosuvastatin | Before Rosuvastatin administration, as well as 30 min, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 h after Rosuvastatin administration

SECONDARY OUTCOMES:
Number of subjects with study drug-related treatment-emergent Adverse Events | Up to 30 days
Area under the concentration-time curve of BAY1841788 from time zero to 24 hours (AUC(0-24)) after single administration | Before BAY1841788 administration, as well as 30 min, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 h after BAY1841788 administration, period 2 day 1
Area under the concentration-time curve of BAY1841788 from time zero to 12 hours (AUC(0-12)) after repeated administration | Before BAY1841788 administration, as well as 30 min, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 h after BAY1841788 administration, period 2 day 7
Maximum drug concentration (Cmax) in plasma of BAY1841788 | Before BAY1841788 administration, as well as 30 min, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 h after BAY1841788 administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Zurth C, Nykanen P, Wilkinson G, Taavitsainen P, Vuorela A, Huang F, Reschke S, Koskinen M. Clinical Pharmacokinetics of the Androgen Receptor Inhibitor Darolutamide in Healthy Subjects and Patients with Hepatic or Renal Impairment. Clin Pharmacokinet. 2022 Apr;61(4):565-575. doi: 10.1007/s40262-021-01078-y. Epub 2021 Dec 6. PMID 34866168